CLINICAL TRIAL: NCT02186717
Title: Does Chewing Gum Hasten Return of Bowel Function Post-operatively in Patients Following Spinal Surgery? A Prospective, Randomized, Controlled Trial
Brief Title: Does Chewing Gum Hasten Return of Bowel Function Post-Operatively in Patients Undergoing Spinal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-065
Record Dates: First submitted 2014-07-02; First posted 2014-07-10 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Return of Bowel Function Following Spinal Surgery
MeSH Terms: interventions — Chewing Gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chewing gum (Experimental): Chewing gum
  Interventions: Dietary Supplement: Chewing gum
- No Chewing Gum (No Intervention): No Chewing Gum

INTERVENTIONS:
Dietary Supplement: Chewing gum — Patients will be asked to chew gum three times a day for 30 minutes each time
  Arms: Chewing gum

SUMMARY:
The specific aim of this prospective, randomized controlled trial is to compare the effect of chewing gum on the return of bowel function in a group of patients undergoing spinal surgery with a group of matched controls that do not receive any chewing gum. A 24-hour reduction in time to passage of first flatus will be considered an important clinical difference.

The research questions are:

1. Does providing chewing gum post-operatively hasten the return of bowel function?
2. Does providing chewing gum post-operatively reduced overall length of stay?
3. Does providing chewing gum post-operatively have any associated complications?
4. Does providing chewing gum post-operatively result in higher objective outcomes scores?

The secondary aims are:

1. To compare hospital length of stay between the groups with a mean of ½ day considered clinically important.
2. To compare time until tolerating regular diet as defined as two consecutive meals with no complications with 24 hours considered statistically significant.
3. To compare incidence and nature of complications between the two groups.
4. To compare the time until completion of rehab milestones with 1 day being considered clinically important.
5. To compare the requirement for nutrition evaluations
6. To compare SF-12 scores as a marker of patient satisfaction with a difference of 10 points or more measured between the two groups upon discharge from hospital and at six-weeks after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Lumbar decompression 2+ levels
* Posterior spinal instrumentation and fusion 1+ levels
* Combined anterior (ALIF/XLIF) and ANY posterior procedure (ie - decompression +/- fusion)

Exclusion Criteria:

* Age < 18
* Trauma
* Tumor
* Infection
* Stand-alone anterior surgery
* Allergy to chewing gum

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2014-06; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Time first pass flatus as a measure of return of bowel function. | Up to two weeks
  Commencing on POD #0 patients will be asked to monitor the time they first pass flatus as a measure of return of bowel function.

SECONDARY OUTCOMES:
length of hospital stay | Up to two weeks
time until tolerating regular diet | Up to two weeks
post-operative narcotic usage | Up to two weeks
pre-operative narcotic usage | Up to two weeks
incidence complications | Up to two weeks
time to completion of rehabilitation criteria for discharge | Up to two weeks
requirement for nutrition evaluations | Up to two weeks
NRS pain scores | Up to two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Russel C. Huang, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No